CLINICAL TRIAL: NCT02996747
Title: Low Grade Chondrosarcoma Versus Enchondroma: Challenges in Diagnosis and Management
Brief Title: Low Grade Chondrosarcoma Versus Enchondroma
Acronym: CONDRO1
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, MD; PhD., Istituto Ortopedico Rizzoli
Other Study IDs: 0016890
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Chondroma; Chondrosarcoma
Keywords: bone tumors; chondroma; chondrosarcoma
MeSH Terms: conditions — Chondroma; Chondrosarcoma; Bone Neoplasms | interventions — Curettage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: curettage (intralesional surgery) — comparison of two different tumors treated by curettage

SUMMARY:
The purpose of this project is to verify possible clinical and radiological findings with regard to distinguishing enchondroma from low grade chondrosarcoma of the long bones. In addition, this study presents the outcome of patients with enchondroma and low grade chondrosarcoma of the long bones who were treated with curettage (intralesional surgery).

DETAILED DESCRIPTION:
The investigators retrospectively review the records of 65 patients with enchondroma and 37 patients with low grade chondrosarcoma of the limbs treated by curettage between 1988 and 2014 in a single Institution.

ELIGIBILITY:
Inclusion Criteria:

* chondroma or low grade chondrosarcoma of long bones

Exclusion Criteria:

* chondroma or low grade chondrosarcoma of spine and pelvis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chondroma or low grade chondrosarcoma of bone treated in a single Institution
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Local recurrence rate of patients with chondroma or low grade chondrosarcoma treated by curettage (intralesional surgery) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Davide Donati, MD, Study Director — Istituto Ortopedico Rizzoli

IPD SHARING:
Plan to Share IPD: Yes
publish a paper in international medical journal